CLINICAL TRIAL: NCT00596154
Title: Rituximab, Methotrexate, Procarbazine and Vincristine Followed by High-dose Chemotherapy With Autologous Stem-cell Rescue in Newly-diagnosed Primary CNS Lymphoma (PCNSL)
Brief Title: Rituximab, Methotrexate, Procarbazine and Vincristine Followed by High-dose Chemotherapy With Autologous Stem-cell Rescue in Newly-diagnosed Primary CNS Lymphoma
Acronym: PCNSL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-129
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-02

CONDITIONS: CNS Lymphoma; CNS Brain Cancer; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Methotrexate; Vincristine; Procarbazine; Busulfan; Thiotepa; Cyclophosphamide; Drug Therapy; Pharmaceutical Preparations

ARMS (1):
- 1 (Experimental): Rituximab, methotrexate (MTX), procarbazine and vincristine (R-MPV). The peripheral blood stem cell (PBSC) harvest procedure will be performed at the discretion of the hematology attending (usually after the 1st or 2nd cycle of R-MPV)and high dose chemotherapy Busulfan, Thiotepa, and Cyclophosphamide. Patients will be off study at the time of death. All patients will be followed for survival every 6 months throughout their lifetime. Survival status may be obtained by phone call, clinical visit or medical records (e.g. physician notes/laboratory results of clinic or hospital visit.
  Interventions: Other: Rituximab, Methotrexate, Vincristine, Procarbazine, PBPCs collection, Busulfan, Thiotepa, and Cyclophosphamide

INTERVENTIONS:
Other: Rituximab, Methotrexate, Vincristine, Procarbazine, PBPCs collection, Busulfan, Thiotepa, and Cyclophosphamide — The initial treatment will consist of cycles of 14 days. Each cycle will start with rituximab, which will be given by vein on day 1.
  On day 2 you will be admitted to the hospital and will receive 3 other drugs:
  Methotrexate will be given by vein over 2 to 3 hours only on day 2. Vincristine will be given as a single injection over a few minutes only on day 2.
  Procarbazine is a pill that you will take at bedtime for 7 nights starting on day 2. Procarbazine is only given every other cycle.
  Other Names: During each cycle, you will receive Rituximab typically as an outpatient on day 1 and then be; admitted on day 2 to receive the other chemotherapy. You will be in the hospital for about 5 days and will be re-admitted to the hospital about 9 days; later to start the next cycle. After each cycle of chemotherapy you will take a medicine called G-CSF to protect you against; infection. PBPCs will be collected when determined by your doctor and may occur with cycle 1 or cycle 2.; You will be admitted again for the high-dose chemotherapy and will receive supportive; medications to help avoid complications, including antibiotics and blood transfusions. Three; drugs, Busulfan, Thiotepa, and Cyclophosphamide will be given to you over 8 days. After a; rest period of approximately 1-2 days, we will give your PBPCs (or bone marrow) back to you; by vein. You will be in the hospital for at least 3 weeks.

SUMMARY:
The purpose of this study is to determine the safety of this new treatment offered in this study. PCNSL can be cured in less than half of patients with standard treatment, a combination of chemotherapy and brain radiation. Also, the combination of chemotherapy and brain radiation may result in serious lasting side effects. Most patients older than age 60 develop memory problems, difficulty walking or inability to control their bladder. Some patients younger than age 60 also develop these side effects.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have non-Hodgkin's lymphoma involving the brain, as demonstrated by CT or MRI and histologic confirmation by one of the following: A positive CSF cytology for lymphoma or a monoclonal lymphocyte population as defined by cell surface markers.

A biopsy of the vitreous or uvea demonstrating non-Hodgkin's lymphoma. Brain biopsy.

* Patients must be HIV-1 negative.
* Patient must have left ventricular ejection fraction ≥ 50%.
* Patients must have no evidence of systemic lymphoma. This must be demonstrated by a CT scan of the chest, abdomen and pelvis prior to registration.
* Patients must have adequate bone marrow function (defined as peripheral leucocyte count >3000 cells/mm3 and platelet count > 100,000 cells/mm3), liver function (bilirubin < 2.0 mg%), and adequate renal function (serum creatinine < 1.5 mg/dl or creatinine clearance > 50cc/min/1.73M2).
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
* Patients must be between 18 and 72 years-old.
* Patients must sign an informed consent.

Exclusion Criteria:

* Prior cranial irradiation
* Other active primary malignancy with the exception of basal cell carcinoma of the skin and cervical carcinoma in situ.
* Pre-existing immunodeficiency such as renal transplant recipient.
* Prior treatment with chemotherapy for CNS lymphoma.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grommes, MD, Principal Investigator — Memorial SloanKettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Omuro A, Correa DD, DeAngelis LM, Moskowitz CH, Matasar MJ, Kaley TJ, Gavrilovic IT, Nolan C, Pentsova E, Grommes CC, Panageas KS, Baser RE, Faivre G, Abrey LE, Sauter CS. R-MPV followed by high-dose chemotherapy with TBC and autologous stem-cell transplant for newly diagnosed primary CNS lymphoma. Blood. 2015 Feb 26;125(9):1403-10. doi: 10.1182/blood-2014-10-604561. Epub 2015 Jan 7. PMID 25568347
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Newly Diagnosed Primary CBS Lymphoma/PCNSL: Rituximab, methotrexate (MTX), procarbazine and vincristine (R-MPV). The peripheral blood stem cell (PBSC) harvest procedure will be performed at the discretion of the hematology attending. Participants will be off study at the time of death.
Period: Overall Study
Arm/Group | Newly Diagnosed Primary CBS Lymphoma/PCNSL
Started | 33
Completed | 31
Not Completed | 2
Not completed — Not Evaluable | 2

BASELINE CHARACTERISTICS:
Arm/Group | Newly Diagnosed Primary CBS Lymphoma/PCNSL
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 57 [24 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated for Toxicity
Description: To evaluate the safety and efficacy of the use of R-MPV followed by high-dose chemotherapy using thiotepa, cyclophosphamide and busulfan with stem cell rescue in patients with newly diagnosed PCSNL.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Diagnosed Primary CBS Lymphoma/PCNSL
Number analyzed (Participants) | 33
Participants | 33

2. Secondary Outcome: Overall Response Rates
Description: To evaluate response rates with the combination of rituximab and MPV as induction chemotherapy.
Time Frame: after 10 weeks (5 cycles)
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Diagnosed Primary CBS Lymphoma/PCNSL
Number analyzed (Participants) | 33
Participants
  Progression Free | 1
  Complete Response | 22
  Partial Response | 6
  Stable Disease | 1
  Not Evaluable | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Newly Diagnosed Primary CBS Lymphoma/PCNSL
All-Cause Mortality (participants affected / at risk) | 7/33
Serious Adverse Events (participants affected / at risk) | 14/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Newly Diagnosed Primary CBS Lymphoma/PCNSL (N=33)
ALT, SGPT (Investigations) | 3
AST, SGOT (Investigations) | 3
Confusion (Psychiatric disorders) | 1
Creatinine (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 2
Fever (in the absence of neutropenia) (General disorders) | 1
Infection, other (Infections and infestations) | 3
Liver dysfunction/failure (Hepatobiliary disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neuropathy: motor (Nervous system disorders) | 1
Obstruction, GI- Small bowel NOS (Gastrointestinal disorders) | 1
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1
Pain - Chest/thorax NOS (General disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Seizure (Nervous system disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Death not related to disease (General disorders) | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Newly Diagnosed Primary CBS Lymphoma/PCNSL (N=33)
Fatigue (General disorders) | 11
Neuropathy: sensory (Nervous system disorders) | 7
Constipation (Gastrointestinal disorders) | 5
Neuropathy: motor (Nervous system disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Lymphopenia (Investigations) | 2
Pain - Head/headache (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT00596154/Prot_SAP_000.pdf